CLINICAL TRIAL: NCT00678730
Title: Pharmacogenetics of Cannabinoid Response
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Principal Investigator, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 0706002754
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: COMT Gene Polymorphism
Keywords: THC; COMT gene polymorphism; schizophrenia; cannabis use
MeSH Terms: conditions — Schizophrenia | interventions — Dronabinol; nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 (Active Comparator): * Very low dose (0.005 mg/kg = 0.35 mg in a 70kg individual) THC, dissolved in ethanol. This dose is roughly equivalent to smoking 1/10th of a marijuana cigarette, or "joint".
  * Low dose (0.025 mg/kg = 1.75 mg in a 70kg individual) THC, dissolved in ethanol. This dose is roughly equivalent to smoking 1/2 of a marijuana cigarette, or "joint".
  * Medium dose (0.05 mg/kg = 3.5 mg in a 70 kg individual) THC, dissolved in ethanol. This dose is roughly equivalent to smoking 1 marijuana cigarette, or "joint".
  Interventions: Drug: delta 9 tetrahydrocannabinol
- 2 (Placebo Comparator): small amount of ethanol, (quarter teaspoon), with no THC
  Interventions: Drug: delta 9 tetrahydrocannabinol

INTERVENTIONS:
Drug: delta 9 tetrahydrocannabinol — 0.05 mg/kg of THC dissolved in ethanol intravenously over 20 minutes
  Other Names: Marijuana; cannabis

SUMMARY:
This study attempts to examine genetic influences on the effects of tetrahydrocannabinol (Δ9-THC), the active ingredient of marijuana, cannabis, "ganja", or "pot".

ELIGIBILITY:
Inclusion Criteria:

* 18 and 55 years (extremes included) on the day of the first dosing.

Exclusion Criteria:

* Cannabis naïve individuals.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2007-08-23 (Actual); Primary Completion 2014-09-11 (Actual); Study Completion 2014-09-11 (Actual)

PRIMARY OUTCOMES:
Behavioral Measures | Baseline, +15, +25, +60, +300

CONTACTS AND LOCATIONS:
Overall Officials: Deepak D'Souza, M.D., Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

REFERENCES:
- [Derived] Ranganathan M, De Aquino JP, Cortes-Briones JA, Radhakrishnan R, Pittman B, Bhakta S, D'Souza DC. Highs and lows of cannabinoid-dopamine interactions: effects of genetic variability and pharmacological modulation of catechol-O-methyl transferase on the acute response to delta-9-tetrahydrocannabinol in humans. Psychopharmacology (Berl). 2019 Nov;236(11):3209-3219. doi: 10.1007/s00213-019-05273-5. Epub 2019 Jun 11. PMID 31187152
- [Derived] Ranganathan M, Radhakrishnan R, Addy PH, Schnakenberg-Martin AM, Williams AH, Carbuto M, Elander J, Pittman B, Andrew Sewell R, Skosnik PD, D'Souza DC. Tetrahydrocannabinol (THC) impairs encoding but not retrieval of verbal information. Prog Neuropsychopharmacol Biol Psychiatry. 2017 Oct 3;79(Pt B):176-183. doi: 10.1016/j.pnpbp.2017.06.019. Epub 2017 Jun 20. PMID 28642081